CLINICAL TRIAL: NCT01783184
Title: Study of Abdominal Aortic Stent Grafts in the Treatment of Infrarenal Abdo Minal Aortic Aneurysms
Brief Title: Study of Abdominal Aortic Stent Grafts in the Treatment of Infrarenal Abdominal Aortic Aneurysms
Status: Completed | Type: Observational
Sponsor: Vascutek Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: EPI-ANA01
Record Dates: First submitted 2013-01-31; First posted 2013-02-04 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

SUMMARY:
The Vascutek Anaconda™ Stent Graft System for repair of Abdominal Aortic Aneurysms (AAA) is the subject of this observational study. 180 patients will be implanted with the Anaconda™ Stent Graft System and will be followed-up annually for 5 years post-implant. The study will satisfy the requirements of the French National Authority for Health (Haute Autorité de santé) and the data collected will be used for reimbursement renewal.

DETAILED DESCRIPTION:
Infrarenal abdominal aortic aneurysms may be treated with the introduction of an abdominal aortic stent graft via the femoral route. This technique is commonly used in high surgical risk patients but can also be suitable under certain conditions for normal risk patients.

Abdominal aortic stent grafts, inserted via the femoral artery, are used to treat infrarenal abdominal aortic aneurysms, removing the need for an invasive surgical procedure.

The aim of this observational study is to evaluate the long-term (5 year) benefits of the technique by documenting the overall mortality, complications (endoleak, migration), rate of surgical conversion, progression and rupture of the aneurysm in a cohort of patients who are representative of the treated population under real conditions of use.

ELIGIBILITY:
Inclusion Criteria:

* Any patient implanted with the Vascutek Anaconda™ Stent Graft System for the treatment of a non-ruptured infrarenal Abdominal Aortic Aneurysm (AAA)

Exclusion Criteria:

* Patients for whom clinical follow-up is impossible and cannot return for check-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Abdominal Aortic Aneurysm (AAA)
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Overall mortality rate | Post-op (within 30 days), 6 months, 12 months and then annually up to 5 years
Mortality rate related to rupture of the aneurysm and relationship to the stent | Post-op (within 30 days), 6 months, 12 months and then annually up to 5 years
Change in diameter of the aneurysm | Post-op (within 30 days), 6 months, 12 months and then annually up to 5 years
Rate of Type I, II and III endoleaks | Post-op (within 30 days), 6 months, 12 months and then annually up to 5 years
Surgical conversion rate | Post-op (within 30 days), 6 months, 12 months and then annually up to 5 years
Rate of endovascular or surgical revisions | Post-op (within 30 days), 6 months, 12 months and then annually up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Professor Dominique Midy, Principal Investigator — Groupe Hospitalier Pellegrin , Bordeaux, France
Locations (26):
- France (26):
  - Clinique Casamance, Aubagne
  - Clinique Saint Etienne, Bayonne
  - Clinique Aguilera, Biarritz
  - Groupe Hospitalier Pellegrin, Bordeaux
  - Centre Hospitalier Jacques Coeur, Bourges
  - C.H. Prive Saint Martin, Caen
  - Infirmerie Protestante, Caluire-et-Cuire
  - Clinique Villette, Dunkirk
  - Centre Hospitalier Universitaire - Hopital Michallon, Grenoble
  - Clinique du Mail, La Rochelle
  - Centre Hospitalier, La Rochelle
  - Hopital Prive de l'Estuaire, Le Havre
  - Clinique de L'Yvette, Longjumeau
  - Clinique Bouchard, Marseille
  - Hopital Fondation Saint Joseph, Marseille
  - Hopital Prive Sainte Blandine, Metz
  - Centre Hospitalier, Moulins
  - Centre Hospitalalier Universitaire - Hopital Brabois, Nancy
  - Polyclinique Francheville, Périgueux
  - Centre Hospitalier, Périgueux
  - Centre Hospitalier de Roanne, Roanne
  - Clinique Saint Hilaire, Rouen
  - Clinique Guillaume de Varye, Saint-Doulchard
  - Clinique de l'Europe, Saint-Nazaire
  - Centre Hospitalier Universitaire - Hopital Civil, Strasbourg
  - Clinique Vauban, Valenciennes

IPD SHARING:
Plan to Share IPD: Undecided